CLINICAL TRIAL: NCT06970054
Title: Home Oscillatory Positive Expiratory Pressure Combined With Aerobic Exercise in Moderate to Severe COPD Patients: A Multicenter, Randomized Controlled Study
Brief Title: Home Oscillatory Positive Expiratory Pressure - Aerobic Exercise Rehabilitation Study
Acronym: HOPE-AERO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: e-Linkcare Meditech Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Huiqing Ge, Director of Respiratory Care Department, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250243
Record Dates: First submitted 2025-04-18; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: COPD; AECOPD
Keywords: Oscillating Positive Expiratory Pressure; OPEP; COPD; AECOPD; Chronic Obstructive Pulmonary Disease; Acute Exacerbation of Chronic Obstructive Pulmonary Disease; Airway Clearance; Global Initiative for Chronic Obstructive Lung Disease; GOLD; aerobic exercise; cardio; COPD management; Internet of Things; IoT
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OPEP only (Experimental): * Patients are provided with an internet-connected handheld respiratory training device.
  * Patients are provided with a wearable device for monitoring data.
  * Patients receive an OPEP training plan and instructions on using the respiratory training device.
  * Training on the OPEP device is conducted:
  * Inpatients: Twice daily training during hospitalization.
  * Outpatients: At least 3 training sessions in the clinic after enrollment.
  * Treatment compliance is monitored remotely via the IoT system for 8 weeks.
  * Patients are scheduled for regular follow-up visits at 1 month, 2 months, 6 months, 12 months, and 24 months (with a window of ±7 days for each visit).
  Interventions: Device: OPEP
- Aerobic Exercise Group (Experimental): * Patients are provided with a wearable device for monitoring data.
  * Patients receive an aerobic exercise training plan and instructions on using the device.
  * Exercise training is conducted:
  * Inpatients: Daily aerobic exercise during hospitalization.
  * Outpatients: At least 3 training sessions in the clinic after enrollment.
  * Treatment compliance is monitored remotely via the IoT system for 8 weeks.
  * Patients are scheduled for regular follow-up visits at 1 month, 2 months, 6 months, 12 months, and 24 months (with a window of ±7 days for each visit).
  Interventions: Behavioral: Aerobic Exercise
- OPEP and Aerobic Exercise (Experimental): * Patients receive both an internet-connected handheld respiratory training device and a wearable device.
  * Patients receive OPEP and aerobic exercise training plans and instructions.
  * Training is conducted:
  * Inpatients: Twice daily OPEP training and daily aerobic exercise during hospitalization.
  * Outpatients: At least 3 training sessions in the clinic after enrollment.
  * Treatment compliance is monitored remotely via the IoT system for 8 weeks.
  * Patients are scheduled for regular follow-up visits at 1 month, 2 months, 6 months, 12 months, and 24 months (with a window of ±7 days for each visit).
  Interventions: Device: OPEP; Behavioral: Aerobic Exercise
- Control (No Intervention): * Patients are advised to maintain their usual activity levels.
  * Patients continue with their prescribed medications.
  * Patients receive routine management, including outpatient education.
  * No specific interventions like respiratory training devices or structured exercise programs are provided.
  * Patients are scheduled for regular follow-up visits at 1 month, 2 months, 6 months, 12 months, and 24 months (with a window of ±7 days for each visit).

INTERVENTIONS:
Device: OPEP — -Patients are provided with a networked handheld respiratory training device. -Patients are provided with a wearable device for monitoring data. -Patients receive an OPEP training plan and instructions on using the respiratory training device. -Training on the OPEP device is conducted: -Inpatients: Twice daily training during hospitalization. -Outpatients: At least 3 training sessions in the clinic after enrollment. -Treatment compliance is monitored remotely via the IoT system for 8 weeks. -Patients are scheduled for regular follow-up visits at 1 month, 2 months, 6 months, 12 months, and 24 months (with a window of ±7 days for each visit).
  Arms: OPEP and Aerobic Exercise; OPEP only
Behavioral: Aerobic Exercise — -Patients are provided with a wearable device for monitoring data. -Patients receive an aerobic exercise training plan and instructions on using the device. -Exercise training is conducted: -Inpatients: Daily aerobic exercise during hospitalization. -Outpatients: At least 3 training sessions in the clinic after enrollment. -Treatment compliance is monitored remotely via the IoT system for 8 weeks. -Patients are scheduled for regular follow-up visits at 1 month, 2 months, 6 months, 12 months, and 24 months (with a window of ±7 days for each visit).
  Arms: Aerobic Exercise Group; OPEP and Aerobic Exercise

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and effectiveness of home OPEP therapy and aerobic exercise training in patients with moderate to severe Chronic Obstructive Pulmonary Disease (COPD) who are at high risk of acute exacerbations, aged 40-80 years. The main questions it aims to answer are:

Does home OPEP therapy, aerobic exercise training, or the combination of both reduce the incidence and hospitalization rate of acute exacerbations of COPD compared to conventional treatment? What are the effects of these interventions on 6-minute walk distance, all-cause mortality, lung function, quality of life, and treatment adherence? Researchers will compare a) conventional treatment, b) OPEP therapy, c) aerobic exercise training, and d) OPEP therapy combined with aerobic exercise training to see if OPEP therapy and/or aerobic exercise training improve pulmonary rehabilitation outcomes.

Participants will:

Receive assigned intervention based on the study arm (conventional treatment, OPEP therapy, aerobic exercise, or combined therapy).

Use respiratory training devices and/or wearable monitoring devices as required by their assigned group.

Follow training plans and therapy schedules. Attend follow-up visits at 1 month, 2 months, 6 months, 12 months, and 24 months.

Complete questionnaires and undergo assessments (e.g., lung function tests, 6-minute walk tests) at baseline and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80 years.
* Diagnosis of AECOPD according to 2025 GOLD criteria, GOLD stage 2-4.
* Patients seeking treatment for acute exacerbation of COPD (AECOPD) as outpatients or inpatients.
* Residing in the study center area with no plans to relocate during the study.
* Voluntary participation with signed informed consent.

Exclusion Criteria:

* Inability to walk or tolerate the 6-minute walk test.
* Inability to cooperate with lung function tests.
* Life expectancy <6 months (e.g., uncontrolled advanced malignancy, recent MI, unstable angina, acute stroke, acute heart failure).
* Active pulmonary tuberculosis or history of lung resection.
* Pregnancy or lactation.
* Liver or kidney failure requiring dialysis.
* Participation in other drug clinical trials or interventional studies.
* Vulnerable populations (e.g., mental illness, cognitive impairment, critically ill, illiterate).
* Other reasons deemed unsuitable by the researcher.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of AECOPD | Over the 24-month follow-up period
  Incidence of moderate to severe acute exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD). Acute exacerbation of COPD is defined according to the Chinese expert consensus on diagnosis and treatment of acute exacerbation of chronic obstructive pulmonary disease (revised edition 2023)
Hospitalization Rates of AECOPD | Over the 24-month follow-up period
  Hospitalization rate of moderate to severe acute exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD). Acute exacerbation of COPD is defined according to the Chinese expert consensus on diagnosis and treatment of acute exacerbation of chronic obstructive pulmonary disease (revised edition 2023)

SECONDARY OUTCOMES:
6-Minute Walk Distance | 1, 2, 6, 12, 24 months, and over 24 months
  Measures the distance a participant can walk in six minutes as an indicator of functional exercise capacity. Higher is better.
All-Cause Mortality | 24 months
Number of Acute Exacerbations | 1, 2, 6, 12, 24 months, and over 24 months
  Total count of acute exacerbation events experienced by each participant.
Proportion of Participants with ≥2 Acute Exacerbations | 24 months
  Percentage of participants experiencing two or more acute exacerbations within 24 months.
Time to First Acute Exacerbation | 24 months
  Duration from study start to the first recorded acute exacerbation for each participant.
COPD Assessment Test (CAT) Score | 1, 2, 6, 12, and 24 months
  Self-reported measure of health status in COPD patients, assessed using the CAT questionnaire. Higher scores indicate a greater impact of COPD on a patient's daily life.
Modified Medical Research Council (mMRC) Dyspnea Score | 1, 2, 6, 12, and 24 months
  Patient-rated scale assessing the severity of breathlessness. Higher grade indicates higher severity.
St. George's Respiratory Questionnaire (SGRQ) Score | 1, 2, 6, 12, and 24 months
  Quality of life assessment specific to respiratory diseases. Higher scores reflect worse health-related quality of life.
Changes in Lung Function Parameter-FVC | 1, 2, 6, 12, and 24 months
  Forced Vital Capacity (FVC) measured in Liters
Changes in Lung Function Parameter-FEV1 | 1, 2, 6, 12, and 24 months
  Forced Expiratory Volume in 1 Second (FEV1) measured in Liters
Changes in Lung Function Parameters - FEV1 predicted | 1, 2, 6, 12, and 24 months
  Predicted Forced Expiratory Volume in 1 second (FEV1 predicted) measured in percentage, calculated using GLI-asian equation
Changes in Lung Function Parameters - FEV1/FVC ratio | 1, 2, 6, 12, and 24 months
  Forced Expiratory Volume in the first second to Forced Vital Capacity (FEV1/FVC ratio), percentage.
Changes in Lung Function Parameters - PEF | 1, 2, 6, 12, and 24 months
  Peak Expiratory Flow (PEF) measured in L/min
Changes in Lung Function Parameters - MMEF | 1, 2, 6, 12, and 24 months
  Maximum Mid-Expiratory Flow (MMEF) percentage of predicted normal
Changes in Blood Gas Parameters - pH | 1, 2, 6, 12, and 24 months
  In arterial blood gas test, pH is a measurement of the acid-base balance of the blood. A normal blood pH range is between 7.35 and 7.45. A pH below 7.35 indicates acidosis, while a pH above 7.45 indicates alkalosis. pH has no units.
Changes in Blood Gas Parameters - PaO2 | 1, 2, 6, 12, and 24 months
  Partial pressure of oxygen (PaO2), in blood gas analysis measures the amount of dissolved oxygen in arterial blood. It's an indicator of oxygenation and is measured in millimeters of mercury (mmHg). A normal PaO2 range is 80-100 mmHg.
Changes in Blood Gas Parameters - PaCO2 | 1, 2, 6, 12, and 24 months
  Partial pressure of carbon dioxide (PaCO2), is a measure of the amount of dissolved carbon dioxide in arterial blood. It's a key indicator of ventilation status, essentially reflecting how well the lungs are removing CO2. It is measured in millimeter mercury (mmHg) and a normal PaCO2 range is 35-45 mmHg.
Changes in Blood Gas Parameters - PaO2/FiO2 | 1, 2, 6, 12, and 24 months
  PaO2/FiO2 ratio is the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction, not a percentage).
Changes in Blood Gas Parameters - HCO3 | 1, 2, 6, 12, and 24 months
  HCO3 refers to the bicarbonate level in the blood, which is a crucial component of acid-base balance. A normal HCO3 range on an ABG is typically between 22 and 26 mEq/L.
Treatment Compliance | 1, 2, 6, 12, and 24 months
  Evaluation of participants' adherence to prescribed treatments and protocols throughout the study using device data and aerobic exercise records.

CONTACTS AND LOCATIONS:
Overall Officials: Huiqing Ge, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bishop JA, Spencer LM, Dwyer TJ, McKeough ZJ, McAnulty A, Alison JA. Changes in Exercise Capacity and Health-Related Quality of Life at Four and Eight Weeks of a Pulmonary Rehabilitation Program in People with COPD. COPD. 2021 Dec;18(6):612-620. doi: 10.1080/15412555.2021.2013793. Epub 2021 Dec 19. PMID 34927525
- [Background] Meghji J, Mortimer K, Agusti A, Allwood BW, Asher I, Bateman ED, Bissell K, Bolton CE, Bush A, Celli B, Chiang CY, Cruz AA, Dinh-Xuan AT, El Sony A, Fong KM, Fujiwara PI, Gaga M, Garcia-Marcos L, Halpin DMG, Hurst JR, Jayasooriya S, Kumar A, Lopez-Varela MV, Masekela R, Mbatchou Ngahane BH, Montes de Oca M, Pearce N, Reddel HK, Salvi S, Singh SJ, Varghese C, Vogelmeier CF, Walker P, Zar HJ, Marks GB. Improving lung health in low-income and middle-income countries: from challenges to solutions. Lancet. 2021 Mar 6;397(10277):928-940. doi: 10.1016/S0140-6736(21)00458-X. Epub 2021 Feb 22. PMID 33631128
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Background] Wang C, Xu J, Yang L, Xu Y, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Huang K, Yao W, Sun T, Shan G, Yang T, Lin Y, Wu S, Zhu J, Wang R, Shi Z, Zhao J, Ye X, Song Y, Wang Q, Zhou Y, Ding L, Yang T, Chen Y, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Chen CS, Wang Z, Zhang H, Bu X, Zhang X, An L, Zhang S, Cao Z, Zhan Q, Yang Y, Cao B, Dai H, Liang L, He J; China Pulmonary Health Study Group. Prevalence and risk factors of chronic obstructive pulmonary disease in China (the China Pulmonary Health [CPH] study): a national cross-sectional study. Lancet. 2018 Apr 28;391(10131):1706-1717. doi: 10.1016/S0140-6736(18)30841-9. Epub 2018 Apr 9. PMID 29650248
- [Background] Celli B, Fabbri L, Criner G, Martinez FJ, Mannino D, Vogelmeier C, Montes de Oca M, Papi A, Sin DD, Han MK, Agusti A. Definition and Nomenclature of Chronic Obstructive Pulmonary Disease: Time for Its Revision. Am J Respir Crit Care Med. 2022 Dec 1;206(11):1317-1325. doi: 10.1164/rccm.202204-0671PP. No abstract available. PMID 35914087
- See also: Global initiative for chronic obstructive lung disease.Global strategy for prevention,diagnosis and management of COPD: 2024 Report — https://goldcopd.org/2024-gold-report/